CLINICAL TRIAL: NCT06659107
Title: Percutaneous Kirschner Wires With Mutual Linking Technique in the Management of Proximal Humeral Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Tony Maher, Lecturer of orthopedic surgery, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: proximal humeral fracture
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Proximal Humeral Fractures
Keywords: Proximal humeral fractures; Mutual linking
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elderly patients with proximal humeral fractures Neer type 2 and 3 (Experimental): Both sexes, age from 60 to 80
  Interventions: Procedure: Closed reduction and fixation by K- wires

INTERVENTIONS:
Procedure: Closed reduction and fixation by K- wires — Fixation by k-wires with mutual linking technique

SUMMARY:
This is study evaluates a novel technique to improve the stability of K-wires used in the fixation of proximal humeral fractures

ELIGIBILITY:
Inclusion Criteria:

* both sexes
* Age from 60 to80 years
* 2 or 3 parts fracture
* recent injury less than 3 weeks

Exclusion Criteria:

* 4 parts fracture
* old injury more than 3 weeks
* previous surgeries or pathologies affecting shoulder range of motion

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
Functional outcome | One year
  Shoulder functional status using the American shoulder and elbow surgeons score (ASES) range from 0 to100, 0 being the worst and 100 being the best
Radiological outcome | 8 weeks
  The percentage of patients achieving union of the fracture assesed by plain X-ray shoulder anteroposterior and lateral views.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No